CLINICAL TRIAL: NCT02021097
Title: A Multicenter, Randomized, Open-labe, Controlled Study to Evaluate the Efficacy and Safety of the Combined Levonorgestrel(LNG) 100mcg and Ethinyl Estradiol(EE) 20mcg for Oral Contraception
Brief Title: Study Evaluating Levonorgestrel and Ethinyl Estradiol for Oral Contraception
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regenex Pharmaceutical, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH-ZQ-03RCT
Record Dates: First submitted 2013-03-12; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Oral Contraceptive
Keywords: Levonorgestrel；; Ethinyl Estradiol；; Oral Contraceptive
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNG100 mcg/EE20 mcg (Experimental)
  Interventions: Drug: Levonorgestrel 100 mcg and Ethinyl Estradiol 20 mcg
- LNG 150mcg/ EE 30mcg (Active Comparator)
  Interventions: Drug: Levonorgestrel 150 mcg and Ethinyl Estradiol 30 mcg

INTERVENTIONS:
Drug: Levonorgestrel 100 mcg and Ethinyl Estradiol 20 mcg — Tablet, orally, opd
  Arms: LNG100 mcg/EE20 mcg
Drug: Levonorgestrel 150 mcg and Ethinyl Estradiol 30 mcg — Tablet, orally, opd
  Arms: LNG 150mcg/ EE 30mcg

SUMMARY:
The purpose of this study is to evaluate the contraceptive efficacy and safety of an oral contraceptive containing a combination of LNG 100mcg/EE 20mcg compared to LNG 150mcg/EE 30 mcg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women,aged 20-35 years who wish to use a contraceptive.
* Women without reproductive system infection complications.
* Willingness to not use other forms of hormonal treatment.
* Three regular menstrual cycles before the study(21-35 days per cycle with 3-7 day's bleeding period, without amenorrhea or irregular bleeding).
* Signed informed consent prior to entry into the trial.

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives.
* Vascular, metabolic, hepatic, renal, oncologic and other diseases.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1008 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy variable is the number of unintended pregnancies as measured by the Pearl Index (PI) during 13 cycles of treatment | From fist dose to 13 treatment cycles (1 cycle=28 days)

SECONDARY OUTCOMES:
Menstrual Cycle Control | From fist dose to 13 treatment cycles (1 cycle=28 days)
  Menstrual cycle control was evaluated by analyzing cycle characteristics, such as cycle length, the incidences of breakthrough bleeding, spotting, and amenorrhea and the duration and intensity of withdrawal bleeding. During the trial, spotting was defined as a light flow that did not necessitate sanitary protection, whereas bleeding was defined as a heavier flow that was similar to normal menstrual flow and necessitated sanitary protection.
Weight changes | From fist dose to 13 treatment cycles (1 cycle=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Chengliang Xiong, Dr, Principal Investigator — Family Planning Research Institute of TJMC,HUST
Locations (17):
- China (17):
  - Beijing, Beijing Municipality
  - Chongqing, Chongqing Municipality
  - Guangzhou, Guangdong
  - Shantou, Guangdong
  - Zhongshan, Guangdong
  - Guiyang, Guizhou
  - Wuhan, Hubei
  - Changde, Hunan
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Yangzhou, Jiangsu
  - Shanghai, Shanghai Municipality
  - Taiyuan, Shanxi
  - Xi’an, Shanxi
  - Tianjin, Tianjin Municipality
  - Ürümqi, Xinjiang
  - Taizhou, Zhejiang